CLINICAL TRIAL: NCT02741518
Title: Fecal Microbiota Transplantation for the Treatment of Obesity
Acronym: FMT Obesity
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Christopher C. Thompson, MD, MSc, Attending Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016P000075
Record Dates: First submitted 2016-04-12; First posted 2016-04-18 (Estimated); Results first posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Obesity
Keywords: obesity; FMT
MeSH Terms: conditions — Obesity | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Active Comparator): The treatment arm will receive an induction dose of FMT via capsules (30) followed by monthly maintenance oral capsules(12) at week 4 and week 8. Donor Stool from healthy lean donors and placebo material will be obtained from OpenBiome. OpenBiome, is a nonprofit 501(c)(3) organization that provides hospitals with screened, filtered, and frozen material ready for clinical use
  Interventions: Biological: Fecal Microbiota Transplantation
- Placebo Arm (Placebo Comparator): The placebo group will receive a placebo FMT capsules at the time of their screening colonoscopy followed by monthly intake of oral placebo capsules at week 4 and week 8
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation — This is pre-screened fecal material that has been encapsulated
  Other Names: FMT
  Arms: Treatment Arm
Other: Placebo — These are capsules that have no fecal material in them.
  Arms: Placebo Arm

SUMMARY:
This is a randomized controlled pilot study to assess the microbiological and clinical impacts of Fecal Microbiota Transplantation (FMT) in patients with obesity. The investigators will prospectively enroll 20 adult patients who are obese (Body Mass Index of 35kg/m2 or higher) after providing written informed consent. The study participants will be randomized 1:1 to either the treatment arm or the placebo arm. The treatment arm will receive an induction FMT with capsules followed by a monthly maintenance dose of oral capsules for 12 weeks total. The placebo group will receive a placebo capsules for induction followed by monthly intake of oral placebo capsules for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Obesity defined as a BMI of 35kg/m2 or higher

Exclusion Criteria:

1. Triglycerides > 500 mg/dL
2. Use of antibiotics <8 weeks prior to participation
3. Use of probiotics <4 weeks prior to participation
4. Alcohol use of greater than 20g/daily or suspicion of alcohol abuse and dependence
5. Substance abuse, current
6. LFTS greater then 3x the ULN
7. Cirrhosis.
8. DM type 2 that is insulin dependent, treated with GLP1-agonists, or poorly controlled on oral medications (HbA1C > 10%)
9. Use of any weight loss medication or participation in a weight loss study or program such as Weight Watchers
10. History of recent weight change (weight loss or weight gain in the two months preceding trial enrollment). This is defined as a gain or loss of 10 or more pounds in the preceding 2 months
11. Patients who are pregnant or breastfeeding
12. Patients who are unable to give informed consent

14. Patients who have previously undergone FMT 15. Patients who have a confirmed malignancy or cancer 16. Patients who are immunocompromised 17. Participation in a clinical trial in the preceding 30 days or simultaneously during this trial 18. Previous gastric or small intestinal surgery that alters gut anatomy such as fundoplication, gastric resection, gastric bypass, small bowel resection, and ileocectomy 19. Other comorbidities including: systemic lupus, inflammatory bowel disease, or Chronic kidney disease as defined by a GFR <60mL/min/1.73m2 44 20. History of rheumatic heart disease, endocarditis, or valvular disease due to risk of bacteremia 21. Any condition, based on clinical judgment that may make study participation unsafe 22. History of severe food allergies 23. Use of immune modulators including methotrexate, mycophenolate mofetil, tacrolimus, cyclosporine, thalidomide, Interleukin-10, or Interleukin-11 24.Treatment with infliximab, adalimumab, certolizumab, natalizumab, vedolizumab or thalidomide 25. Congenital or acquired immunodeficiencies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2019-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C Thompson, MD, MSC, Principal Investigator — Brigham and Women's Hospital; Jessica R Allegretti, MD, MPH, Study Director — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Allegretti JR, Kassam Z, Hurtado J, Marchesi JR, Mullish BH, Chiang A, Thompson CC, Cummings BP. Impact of fecal microbiota transplantation with capsules on the prevention of metabolic syndrome among patients with obesity. Hormones (Athens). 2021 Mar;20(1):209-211. doi: 10.1007/s42000-020-00265-z. Epub 2021 Jan 9. PMID 33420959
- [Derived] Allegretti JR, Kassam Z, Mullish BH, Chiang A, Carrellas M, Hurtado J, Marchesi JR, McDonald JAK, Pechlivanis A, Barker GF, Miguens Blanco J, Garcia-Perez I, Wong WF, Gerardin Y, Silverstein M, Kennedy K, Thompson C. Effects of Fecal Microbiota Transplantation With Oral Capsules in Obese Patients. Clin Gastroenterol Hepatol. 2020 Apr;18(4):855-863.e2. doi: 10.1016/j.cgh.2019.07.006. Epub 2019 Jul 10. PMID 31301451

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm | Placebo Arm
Started | 11 | 11
Completed | 10 | 10
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Placebo Arm | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Full Range); unit: years] | 44.5 [18 to 63] | 43.3 [25 to 65] | 43.9 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 9 | 11 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 11 | 22
BMI [Mean (Full Range); unit: Kg/m^2] | 41.1 [35 to 51.7] | 40.4 [36 to 49.1] | 40.8 [35 to 51.7]

OUTCOME MEASURES:

1. Primary Outcome: Adverse Event Frequency
Description: Number of patients reporting adverse events
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 11 | 11
Participants
  Patients experiencing AEs | 11 | 11
  Patients who Experienced SAE | 1 | 0

2. Secondary Outcome: Assess Change of AUC of GLP-1 as a Therapeutic Biomarker for Clinical Response to Fecal Microbiota Transplantation From Baseline to Week 12
Description: Fecal Microbiota Transplantation will lead to an increase in short chain fatty acids which will lead to an increase in the metabolic regulator GLP-1
Time Frame: 12 weeks
Population: Population analyzed includes all subjects except for the two subjects who withdrew mid study
Measure: Mean (Standard Error); unit: pg/ml x minutes
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 10 | 10
pg/ml x minutes | 509.6 (318.7) | 311.3 (261)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course 6 months
Arm/Group | Treatment Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/11
Other Adverse Events (participants affected / at risk) | 11/11 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=11) | Placebo Arm (N=11)
ER Visit for Vomiting and Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Post final FMT dose patient experienced an episode of Diarrhea and 4 episodes of vomiting. They proceeded to the ER where they were determined to be afebrile. Labs were all within normal limits and ER reported subject drinking un-pasteurized milk.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=11) | Placebo Arm (N=11)
Bloating (Gastrointestinal disorders) | 3 (4) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 5 (6) | 7 (13)
Diarrhea (Gastrointestinal disorders) | 6 (9) | 6 (8)
Blood in stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gas (Gastrointestinal disorders) | 1 (1) | 2 (2)
Heartburn (Gastrointestinal disorders) | 1 (2) | 1 (1)
Insect Bite (General disorders) | 1 (1) | 0 (0)
Bruises (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 1 (1)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 2 (3) | 2 (2)
Nausea (General disorders) | 3 (6) | 1 (1)
Vomiting (General disorders) | 1 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT02741518/Prot_SAP_000.pdf